CLINICAL TRIAL: NCT06003907
Title: Effectiveness of Graston and Cupping Applications in Individuals With Cervical Disc Herniation: A Randomized Controlled Trial
Brief Title: Comparison of Conservative Treatment and Graston and Cup Applications in Patients With Cervical Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar65
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain; Cervical Disc Herniation
Keywords: graston technique; cupping therapy
MeSH Terms: conditions — Neck Pain | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: conservative and traditional physiotherapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physiotherapy (Active Comparator): traditional and complementary medicine methods will not be used.
  Interventions: Other: conventional
- cupping therapy and graston (Experimental): Complementary methods will be used alongside conventional physiotherapy.
  Interventions: Other: conventional; Other: traditional and complementary medicine methods

INTERVENTIONS:
Other: conventional — hot application electrotherapy ultrasound mobilization joint range of motion exercises stretching exercises balance exercises posture exercises
Other: traditional and complementary medicine methods — The Graston Technique is a form of manual therapy known as instrument assisted soft tissue mobilization. Graston massage is performed using titanium-coated metal rods specially designed for different parts of the body.
  Cupping therapy is a treatment method that creates a regional vacuum to increase the blood circulation of the person and provide healing.
  Arms: cupping therapy and graston

SUMMARY:
The aim of the study is to examine the effects of graston and dry cupping techniques applied in addition to the conservative treatment program on neck awareness, grip strength, balance and sleep quality in patients with cervical disc herniation between the ages of 18-65.

DETAILED DESCRIPTION:
The research will be carried out on 30 cases diagnosed with cervical disc herniation between the ages of 18-65. The patients will be divided into 2 groups as control and experimental groups by simple randomization method. While the conservative physical therapy program is applied to the control group, the patients in the experimental group will be applied 1 day graston and 1 day dry cup technique in addition to the ones in the experimental group. All patients will be treated for 20 sessions, 5 days / 4 weeks. Fremantle Neck Awareness Questionnaire to assess neck awareness, hand dynamometer to assess grip strength, Berg Balance Scale to assess balance and Jenkins Sleep Scale to assess sleep quality will be used. All tests will be measured at the start of treatment and after 4 weeks of intervention. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being diagnosed with cervical disc herniation
* Being diagnosed with cervical disc herniation at the level of bulging or protrusion according to MRI results

Exclusion Criteria:

* Presence of cervical spine surgery history
* Presence of primary or spinal metastatic malignancy
* Having vascular problems
* Individuals with sleep apnea
* Those who use psychiatric drugs
* Presence of various pathologies in the upper extremity (fracture, ganglion cyst, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
The Fremantle Neck Awareness Questionnaire | 6 weeks
  It is a 9-question questionnaire that evaluates the way people perceive the communication between their neck and their body, and the way they perceive their body position. Evaluates the perception that differs according to the individual. It is a Likert-type questionnaire (0 = Never/Never feel this way, 1= I rarely feel this way, 2 = Sometimes, or sometimes I feel this way, 3 = I feel this way often, 4 = I feel this way all or most of the time)
Berg Balance Scale | 6 weeks
  The Berg Balance Scale is a scale developed for the assessment of postural control in adults and is easily used in many areas of rehabilitation. It consists of 14 items in total. Scoring evaluates whether the patient can safely perform a task in a given amount of time. High fall risk and balance disorder between 0-20 points; A score of 21-40 indicates moderate risk of falling and an acceptable balance; A score of 41 and above indicates good balance and minimal risk of falling.
Jenkins Sleep Scale | 6 weeks
  The Jenkins Sleep Scale is used in clinical studies to evaluate the sleep problems of patients. Patients are asked 4 questions about sleep problems in the last month and are asked to answer them. 0 (hardly), 1 (1-3 days per month), 2 (4-7 days per month), 3 (8-14 days per month), 4 (15-21 days per month), 5 (23-31 days per month)

CONTACTS AND LOCATIONS:
Overall Officials: Beste İNCEKULAK, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keramat KU, Gaughran A. Safe physiotherapy interventions in large cervical disc herniations. BMJ Case Rep. 2012 Aug 18;2012:bcr2012006864. doi: 10.1136/bcr-2012-006864. PMID 22907861
- [Background] Crothers A, Walker B, French SD. Spinal manipulative therapy versus Graston Technique in the treatment of non-specific thoracic spine pain: design of a randomised controlled trial. Chiropr Osteopat. 2008 Oct 30;16:12. doi: 10.1186/1746-1340-16-12. PMID 18959807
- [Background] Choi TY, Ang L, Ku B, Jun JH, Lee MS. Evidence Map of Cupping Therapy. J Clin Med. 2021 Apr 17;10(8):1750. doi: 10.3390/jcm10081750. PMID 33920643
- [Background] Kim S, Lee SH, Kim MR, Kim EJ, Hwang DS, Lee J, Shin JS, Ha IH, Lee YJ. Is cupping therapy effective in patients with neck pain? A systematic review and meta-analysis. BMJ Open. 2018 Nov 5;8(11):e021070. doi: 10.1136/bmjopen-2017-021070. PMID 30397006
- [Background] Abdel-Aal NM, Elsayyad MM, Megahed AA. Short-term effect of adding Graston technique to exercise program in treatment of patients with cervicogenic headache: a single-blinded, randomized controlled trial. Eur J Phys Rehabil Med. 2021 Oct;57(5):758-766. doi: 10.23736/S1973-9087.21.06595-3. Epub 2021 May 5. PMID 33947825